CLINICAL TRIAL: NCT05414357
Title: Impact of Sleep Disturbance on Cognition and Quality of Life in Breast Cancer
Acronym: ICANSLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: UMR_S 1077 Inserm-EPHE-Normandie Université (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A00437-36
Record Dates: First submitted 2022-05-30; First posted 2022-06-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Sleep; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with chemotherapy (Experimental)
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging at rest and in activation with attentional task
- Patients without chemotherapy (Active Comparator)
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging at rest and in activation with attentional task
- cancer-free volunteers (Active Comparator)
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging at rest and in activation with attentional task

INTERVENTIONS:
Diagnostic Test: Functional Magnetic Resonance Imaging at rest and in activation with attentional task — Participants complete 3 successive assessments (T1: baseline, T2: at 6 months, T3: after galvanic vestibular stimulation). Assessments include:
  * Functional and Anatomic Magnetic Resonance Imaging at rest and in activation (only at T1 and T2).
  * Biological and physiological measurements
  * Spatial memory task
  * Cognitive battery
  * Questionnaires (sleep, quality of life)
  Other Names: Spatial memory task; Cognitive battery; quality of life questionnaires

SUMMARY:
Patients treated for breast cancer frequently complain of sleep disturbances, about 40% of them. Of the sleep disturbances experienced by patients, insomnia is the most common complaint. The prevalence of insomnia complaints is higher in breast cancer patients compared to other types of cancer, and is also higher than in the general population (between 20% and 70% in breast cancer patients vs 30% in the general population). A recent study indicates that sleep complaints concern 25% of patients even before diagnosis, and 46% (including 18% complaining of insomnia) at the time of diagnosis, showing the negative impact of the announcement of the pathology on the subjective quality of sleep, and particularly on symptoms suggestive of insomnia. However, objective information on a modification of sleep patterns in breast cancer remains scarce and does not allow us to conclude. In particular, previous studies have focused only on the effects of chemotherapy and have not always included a control group, limiting the significance of their results. The links with cognitive and psychopathological processes and the underlying mechanisms are not clearly demonstrated in this pathology. Finally, taking into account patients' complaints, it appears necessary to limit sleep disorders in breast cancer in order to improve patients' quality of life using non-medicinal and easy-to-implement approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 39 to 69 years
* Patient with operated localized breast cancer who may or may not be starting adjuvant chemotherapy
* Patient with education level 3 "end of primary education"
* Patient with a good command of the French language
* Patient with access to the Internet from a computer at home
* Patient having signed the consent to participate in the study
* Patient with no pre-existing cognitive impairment at the time of cancer diagnosis
* Patient with a sleep complaint (ISI > 7)

Exclusion Criteria:

* Patient with metastatic cancer
* Patient with a primary cancer other than breast cancer
* Patient with a history of neurological damage
* Patient with treated sleep apnea
* Patient with drug use or alcohol abuse (≥3 drinks/day on average and/or >10 drinks/week)
* Patient with a treatment that has not been stabilized for at least 3 months (hypnotics, antidepressants, anxiolytics)
* Patient with a personality disorder and/or an evolving psychiatric pathology
* Patient with a contraindication to MRI (claustrophobia, metallic objects in the body)
* Patient with an uncorrected vision problem

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Ratio of total sleep time to time spent in bed and the number of awakenings lasting more than one minute measured by polysomnography with actimeter | At 6 months
Amplitude of activity-rest rhythm measured with actimeter | At 6 months
Acrophase of activity-rest rhythm measured with actimeter | At 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Inserm-Ephe-Unicaen U1077, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galin M, de Girolamo L, Clarisse B, Segura-Djezzar C, Glockner F, Elia C, Rehel S, Clochon P, Doidy F, Chavant J, Etard O, Viader F, Grellard JM, Lequesne J, Joly F, Eustache F, Martin T, Giffard B, Quarck G, Perrier J. Exploration of effects of galvanic vestibular stimulation on circadian rhythms and its associations with sleep and spatial memory in patients with breast cancer: The ICANSLEEP-2 protocol. PLoS One. 2024 Jul 31;19(7):e0306462. doi: 10.1371/journal.pone.0306462. eCollection 2024. PMID 39083526
- [Derived] Elia C, de Girolamo L, Clarisse B, Galin M, Rehel S, Clochon P, Doidy F, Segobin S, Viader F, Naveau M, Delcroix N, Segura-Djezzar C, Grellard JM, Lequesne J, Etard O, Martin T, Quarck G, Eustache F, Joly F, Giffard B, Perrier J. Effects of sleep disturbances and circadian rhythms modifications on cognition in breast cancer women before and after adjuvant chemotherapy: the ICANSLEEP-1 protocol. BMC Cancer. 2023 Dec 1;23(1):1178. doi: 10.1186/s12885-023-11664-x. PMID 38041077